CLINICAL TRIAL: NCT05779631
Title: Multi-parametric MRI in Patients Suspected for Muscle Invasive Bladder Cancer: a New Local Staging Paradigm (BladParadigm)
Brief Title: Multi-parametric MRI in Patients Suspected for Muscle Invasive Bladder Cancer: a New Local Staging Paradigm
Acronym: BladParadigm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-15859
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer; Muscle-invasive Bladder Cancer
Keywords: mpMRI + same-day biopsy; TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: TURBT versus mpMRI plus a same-day cystoscopic bladder biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mpMRI plus a same-day cystoscopic bladder biopsy (Experimental): multiparametric MRI plus same-day cystoscopic bladder biopsy
  Interventions: Diagnostic Test: mpMRI plus a same-day cystoscopic bladder biopsy
- TURBT (Active Comparator): Transurethral resection of the bladder tumor, blood withdrawal shortly before and after TURBT
  Interventions: Procedure: TURBT

INTERVENTIONS:
Diagnostic Test: mpMRI plus a same-day cystoscopic bladder biopsy — mpMRI plus a same-day cystoscopic bladder biopsy
  Arms: mpMRI plus a same-day cystoscopic bladder biopsy
Procedure: TURBT — Transurethral resection of the bladder tumor, blood withdrawal shortly before and after TURBT
  Arms: TURBT

SUMMARY:
A two-arm multicenter randomised controlled trial, comparing progression free survival, time to definitive treatment and cost-effectiveness of the standard of care (TURBT) and mpMRI followed by same-day cystoscopic bladder biopsy for diagnosis of patients with suspicion of muscle-invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18+ years of age)
* Clinically suspected MIBC
* No lymph node or distant metastases
* Written informed consent

Exclusion Criteria:

* Unable or unwilling to undergo mpMRI
* Unfit for TURBT
* Unfit for definitive treatment with curative intent
* A history of cancer, including bladder cancer, except: non-melanoma skin cancer, prostate cancer on active surveillance or a solid malignant tumor ≥5 years disease-free since last treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Progression-free survival, defined as the time between randomisation and one of the following events, whichever occurs first:
  * Diagnosis of distant metastases
  * Diagnosis of loco-regional nodal recurrence
  * Death from any cause

SECONDARY OUTCOMES:
Time to definitive treatment | 2 years
  Definitive treatment is defined as TURBT in case of NMIBC and radical cystectomy with or without neoadjuvant chemotherapy or chemoradiotherapy in case of MIBC. Time to definitive treatment is the time between randomisation and the first of these mentioned treatments.
Health-related quality of life | 2 years
  Generic health-related quality of life will be assessed at baseline, 6 months, 12 months and 24 months using the EuroQol 5 dimensions 5 levels (EuroQol 5D) questionnaire.
Hospital-related healthcare costs | 2 years
  Hospital registries will be used to identify all items / procedures / activities related to the management of the bladder cancer and obtain a valid and reliable estimate of the costs. Unit costs will be based on the Dutch manual for costing studies.
Cost-effectiveness | 2 years
  Unit costs will be based on the Dutch manual for costing studies. Effectiveness will be measured in terms of quality-adjusted life years (QALYs), following the Dutch guideline for economic evaluation (EuroQol 5D).
Circulating tumor cells | Before (at least on same day) and after (max. 60 minutes) TURBT
  Percentage of patients with CTCs/CTC clusters in the blood sample post-TURBT, among those who were CTC-free pre-TURBT, analysed by blood withdrawal shortly before and after TURBT.
Metastatic potential of CTC-positive samples | Before (at least on same day) and after (max. 60 minutes) TURBT
  Post-TURBT CTC-positive samples of patients that were CTC negative prior to TURBT will be further analyzed for the expression levels of bladder cancer metastasis-associated genes using principal component- and heatmap analysis.

CONTACTS AND LOCATIONS:
Overall Officials: A. G. van der Heijden, Dr., Principal Investigator — Radboud University Medical Center
Locations (19):
- Netherlands (19):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Ziekenhuisgroep Twente, Almelo
  - Meander MC, Amersfoort
  - Amsterdam UMC, location AMC, Amsterdam
  - Amsterdam UMC, location VUmc, Amsterdam
  - Antoni van Leeuwenhoek - Netherlands Cancer Institute, Amsterdam
  - OLVG, Amsterdam
  - Rijnstate ziekenhuis, Arnhem
  - Maasziekenhuis Pantein, Boxmeer
  - Ziekenhuis Gelderse Vallei, Ede
  - Treant, Emmen
  - Medisch Spectrum Twente, Enschede
  - St. Antonius ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud university medical center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Bernhoven ziekenhuis, Uden
  - University Medical Center Utrecht, Utrecht
  - VieCuri medisch centrum, Venlo

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data are available upon request to other research groups
Supporting Information: Study Protocol, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] van Koeverden SW, van Hoogstraten LM, de Rooij M, van der Leest M, Grutters JP; BladParadigm study group; Kiemeney LA, van der Heijden AG. Multiparametric MRI for local staging in patients with suspected muscle-invasive bladder cancer: study protocol for a multicentre, non-inferiority randomised controlled trial (the BladParadigm study). BMJ Open. 2025 Aug 16;15(8):e100002. doi: 10.1136/bmjopen-2025-100002. PMID 40819867